CLINICAL TRIAL: NCT02819037
Title: Modification of Digestive Flora After Gastric Bypass : Pilot Study on Microbial Overgrowth Using Gas Chromatography
Brief Title: Small Intestinal Bacterial Overgrowth Obese
Acronym: SIBOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: Santelys Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0046; 2015-A01807-42 (Other: ANSM)
Record Dates: First submitted 2016-06-21; First posted 2016-06-30 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Gastric Bypass; Blind Loop Syndrome; Bacterial Overgrowth Syndrome; Chromatography, Gas
Keywords: Gastric bypass; Intestinal Bacterial Overgrowth Syndrome; Gas chromatography
MeSH Terms: conditions — Blind Loop Syndrome; Mucopolysaccharidosis IV | interventions — Chromatography, Gas; Occult Blood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gas chromatography and stool analysis (Experimental): gas chromatography and stool analysis for detection of malabsorption
  Interventions: Procedure: gas chromatography; Procedure: Stool analysis for detection of malabsorption

INTERVENTIONS:
Procedure: gas chromatography
Procedure: Stool analysis for detection of malabsorption

SUMMARY:
The objective of this research is to determine the incidence of microbial overgrowth of the small intestine before and after a gastric bypass. For this purpose, the study is based on the analysis of the expired hydrogen H2 with gas chromatography before surgery and at 1, 3, 6, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Severe obesity (BMI>35kg/m² with at least one comorbidity or BMI>40kg/m² without comorbidity) and after medical care for at least 6 months
* Patient who will follow bariatric surgery by bypass gastric
* Social insurance affiliation
* Signature of the informed consent

Exclusion Criteria:

* Contraindication criteria for bariatric surgery (cognitive or mental severe disorders, severe and non-stabilized eating disorders, etc.)
* Chronic inflammatory bowel disease (Crohn's disease, hemorrhagic rectocolitis)
* Previous intestinal surgery
* Antibiotic periodicity treatment of less than 3 months
* Other diseases responsible for bacterial overgrowth
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Changes in expired hydrogen H2 concentration | change at baseline et up to 24 months
  Measured by gas chromatography

SECONDARY OUTCOMES:
Changes in digestive symptoms | change at baseline et up to 24 months
Changes in intestinal transit | change at baseline et up to 24 months
  Characterisation of intestinal transit by measuring stool frequency
Changes in malabsorption | change at baseline et up to 24 months
  Detection of lipids, vitamins (A, B1, B9, B12, D, E), zinc, magnesium, phosphorus, serum iron and protein balance (albumin, prealbumin, CRP) in order to diagnosis the presence of malabsorption

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Florent, MD, PhD, Study Director — Centre Hospitalier Arras
Locations (2):
- France (2):
  - Centre Hospitalier d'Arras, Arras
  - Centre Hospitalier de Douai, Douai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Florent V, Dennetiere S, Gaudrat B, Andrieux S, Mulliez E, Norberciak L, Jacquez K. Prospective Monitoring of Small Intestinal Bacterial Overgrowth After Gastric Bypass: Clinical, Biological, and Gas Chromatographic Aspects. Obes Surg. 2024 Mar;34(3):947-958. doi: 10.1007/s11695-024-07080-0. Epub 2024 Feb 1. PMID 38300481